CLINICAL TRIAL: NCT00274768
Title: Phase II Study of Fixed-Dose Capecitabine in Metastatic Breast Cancer
Brief Title: Capecitabine in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0425 CDR0000446286; P30CA006973 (NIH); JHOC-J0425 (Other: SKCCC); JHOC-SKCCC-J0425 (Other: SKCCC); JHOC-IRB-04032502 (Other: SKCCC)
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Results first posted 2012-12-21 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; male breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Capecitabine (Experimental): 26 patients received the pre-defined starting dose of capecitabine of 3,000 mg orally daily given in two divided doses. Two thirds of the patients received either the same dose or a 500 mg lower dose compared to what would have been administered with a commonly used body surface area (BSA)-dosing schedule (2,000 mg/m2 with rounding down to nearest 500 mg multiple).
  Interventions: Drug: capecitabine

INTERVENTIONS:
Drug: capecitabine — A total of 115 cycles of therapy were administered and five patients did not complete cycle 1. The median number of cycles initiated was four (range 1-16).
  Other Names: Xeloda

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well capecitabine works in treating patients with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with metastatic breast cancer treated with a fixed-dose of capecitabine.

Secondary

* Determine the clinical benefit, time to treatment failure (TTF), safety, and toxicity profile of this regimen in these patients.
* Determine the pharmacokinetics (PK) and pharmacogenetics in these patients.
* Correlate pharmacodynamic effects of this drug with toxicity and response in these patients.
* Determine compliance and adherence to this regimen and correlate with PK parameters in these patients.

OUTLINE: This is an open-label study.

Patients receive a fixed-dose of oral capecitabine twice daily on days 1-14. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically.

PROJECTED ACCRUAL: A total of 45 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of adenocarcinoma of the breast

  * Evidence of metastatic involvement (stage IV disease)
* Patients must have measurable disease

  * At least one measurable lesion as defined by the Response Evaluation Criteria in Solid Tumors (RECIST)
* Treated brain metastases (surgery or radiation therapy) allowed if clinically stable
* Patients with leptomeningeal disease are ineligible
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Male or female
* Menopausal status not specified
* Absolute neutrophil count (ANC) ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Creatinine clearance > 50 mL/min
* Fertile patients must use effective contraception
* No history of another severe and/or life-threatening medical disease
* No other active primary malignancy
* Not pregnant or nursing
* Negative pregnancy test
* Patients with asymptomatic HIV infection are eligible
* Liver dysfunction score ≤ 9
* No pre-existing liver disease (i.e., cirrhosis or active viral hepatitis)
* No active gastrointestinal malabsorption illness
* No clinically significant cardiac disease, including the following:

  * Congestive heart failure, symptomatic coronary artery disease, and cardiac arrhythmias not well controlled with medication, or myocardial infarction within the past six months
* No prior unanticipated severe reaction to fluoropyrimidine therapy, known hypersensitivity to fluorouracil, or known dihydropyrimidine dehydrogenase deficiency
* No history of uncontrolled seizures or central nervous system disorders
* No significant history of noncompliance to medical regimens
* No clinically significant psychiatric disability that would preclude study compliance

PRIOR CONCURRENT THERAPY:

* No previous capecitabine
* Up to 3 prior cytotoxic regimens allowed for metastatic disease

  * Prior noncytotoxic therapy allowed (e.g., hormonal treatment or trastuzumab)
* No other concurrent therapies intended to treat the primary condition including chemotherapy, biologic agents, or immunotherapy
* No concurrent anti-estrogen therapy, radiation therapy, or investigational systemic therapy
* No other concurrent investigational drugs
* No concurrent use of the following drugs: warfarin for full anticoagulation, cimetidine, or azidothymidine (AZT)

  * Mini-dose warfarin for prophylaxis of central venous catheter thrombosis allowed
* At least 4 weeks since prior sorivudine or brivudine
* Concurrent use of bisphosphonates allowed if initiated before beginning study therapy
* Concurrent use of megestrol acetate suspension as an appetite stimulant allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-04; Primary Completion 2009-12 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C. Wolff, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (3):
- United States (3):
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Fackler MJ, Lopez Bujanda Z, Umbricht C, Teo WW, Cho S, Zhang Z, Visvanathan K, Jeter S, Argani P, Wang C, Lyman JP, de Brot M, Ingle JN, Boughey J, McGuire K, King TA, Carey LA, Cope L, Wolff AC, Sukumar S. Novel methylated biomarkers and a robust assay to detect circulating tumor DNA in metastatic breast cancer. Cancer Res. 2014 Apr 15;74(8):2160-70. doi: 10.1158/0008-5472.CAN-13-3392. PMID 24737128

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty patients with metastatic breast cancer were consented between August 2005 and December 2008. Twenty six patients were eligible and initiated treatment on-study.
Pre-assignment Details: Women (≥ 18 or older) with a histologically confirmed metastatic (stage 4) adenocarcinoma of the breast were eligible. Several inclusion and exclusion applied to confirm that women were appropriate to take part in the study intervention.
Groups:
- Capecitabine: The starting dose of capecitabine was 3,000 mg (total daily dose) given in two divided daily doses for 14 days followed by 7 days of rest (1 cycle = 21 days). Missed doses were not substituted. Treatment was continued until unacceptable toxicity, disease progression, or withdrawal of consent.
Period: Overall Study
Arm/Group | Capecitabine
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Capecitabine
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT/MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Participants were followed to progression, evaluated every 12 weeks
Population: Any participant who completed at least one (1) cycle of capecitabine administration was evaluable for response.
Measure: Number; unit: participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 21
participants | 21

2. Secondary Outcome: Clinical Benefit as Assessed by Lack of Progression for at Least 24 Weeks
Description: The overall clinical benefit rate as assessed by number of participants with lack of progression for at least 24 weeks.
Time Frame: 3-week cycles of treatment up to 16 cycles
Population: Five patients did not complete cycle 1
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 21
Participants | 4

3. Secondary Outcome: Pharmacokinetics of Capecitabine and Metabolites as Assessed by Maximum Plasma Concentration
Description: Pharmacokinetics of Capecitabine and metabolites [5-fluoro-5'-deoxycytidine (5'-DFCR), 5-fluoro-5'-dexoxyuridine (5'-DFUR), and 5-fluorouracil (FU)] assessed using maximum plasma concentration (Cmax) in ng/mL.
Time Frame: 0.25, 0.5, 1, 2, 3, 4, 5, 6 and 8 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Capecitabine
Number analyzed (Participants) | 26
ng/mL
  Capecitabine | 9324 (7015)
  5'-DFCR | 6353 (2590)
  5'-DFUR | 4597 (2608)
  5-FU | 753 (1209)

4. Secondary Outcome: Pharmacokinetics of Capecitabine and Metabolites as Assessed by Area Under the Curve (AUC)
Description: Pharmacokinetics of Capecitabine and metabolites [5-fluoro-5'-deoxycytidine (5'-DFCR), 5-fluoro-5'-dexoxyuridine (5'-DFUR), and 5-FU] assessed using AUC in ng*h/mL.
Time Frame: 0.25, 0.5, 1, 2, 3, 4, 5, 6 and 8 hours
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Capecitabine
Number analyzed (Participants) | 26
ng*h/mL
  Capecitabine | 7255 (4180)
  5'-DFCR | 11344 (5583)
  5'-DFUR | 6653 (2166)
  5-FU | 1230 (1826)

5. Secondary Outcome: Adherence and Compliance to Oral Medication Using Electronic Monitoring
Description: This was assessed by number of participants who did not miss any doses of Capecitabine during treatment using the Medication Event Monitoring System (MEMS).
Time Frame: 3-week cycles of treatment up to 16 cycles
Measure: Count of Participants; unit: Participants
Arm/Group | Capecitabine
Number analyzed (Participants) | 26
Participants | 13

6. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure in weeks
Time Frame: 3-week cycles of treatment up to 16 cycles
Population: Five patients did not complete cycle 1
Measure: Median (Full Range); unit: weeks
Arm/Group | Capecitabine
Number analyzed (Participants) | 21
weeks | 12 [6 to 48]

ADVERSE EVENTS:
Time Frame: Participants were evaluated for adverse events every cycle, or every 3 weeks; median length of time on trial was 7 cycles (or 21 weeks). Potentially treatment-related toxicities of all grades and for all cycles are listed.
Arm/Group | Capecitabine
All-Cause Mortality (participants affected / at risk) | 2/26
Serious Adverse Events (participants affected / at risk) | 2/26
Other Adverse Events (participants affected / at risk) | 20/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine (N=26)
Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) — Participant death due to rapid progression of metastatic breast cancer; not related to study intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Capecitabine (N=26)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Fatigue (General disorders) | 16 (16)
Anorexia (Metabolism and nutrition disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 14 (14)
Vomiting (General disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Constipation (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 6 (6)
Dysgeusia (Nervous system disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 20 (20)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The small sample size limited a number of the secondary objectives.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No